CLINICAL TRIAL: NCT05240131
Title: An Open Label Study Followed by a Randomised, Double-blind, Placebo-controlled, Parallel Group and an Extension Study to Investigate the Safety and Efficacy of GB1211 (a Galectin-3 Inhibitor) in Combination With Atezolizumab in Patients With Non-Small Cell Lung Cancer (NSCLC).
Brief Title: A Study to Investigate the Safety and Efficacy of GB1211 (a Galectin-3 Inhibitor) in Combination With Atezolizumab in Patients With Non-Small Cell Lung Cancer (NSCLC).
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Collaborators: Linical Europe GmbH (Unknown); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GALLANT-1
Record Dates: First submitted 2022-01-27; First posted 2022-02-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Part A is an open label dose ascending design. PART B is a randomised, double-blind, placebo-controlled, parallel group design PART C is an extension study to assess long-term safety and tolerability
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PART A open label PART B & C will be double blind until the primary analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A - GB1211 200 mg and 100 mg BID in combination with atezolizumab. (Experimental): Part A of the study, open-label sentinel dosing will be undertaken to assess safety and tolerability of GB1211 at 200 mg and 100 mg BID in combination with atezolizumab.
  Interventions: Drug: GB1211; Drug: Atezolizumab
- Part B - GB1211 (200 or 100 mg BID) or Placebo in addition to atezolizumab (Experimental): Part B of the study, GB1211 (200 or 100 mg BID to be selected from part A) in addition to atezolizumab, for 12 weeks
  Interventions: Drug: GB1211; Drug: Placebo; Drug: Atezolizumab
- Part C - Extension of GB1211 (200 or 100 mg BID) or Placebo in addition to atezolizumab (Experimental): Extension of GB1211 in addition to atezolizumab until part B has been unblinded.
  Extension of placebo in addition to atezolizumab until part B has been unblinded
  Interventions: Drug: GB1211; Drug: Placebo; Drug: Atezolizumab

INTERVENTIONS:
Drug: GB1211 — GB1211 is a galectin 3 inhibitor an orally available small molecular anti-fibrotic. It is administered orally twice a day.
Drug: Placebo — Placebo is administered orally twice a day.
  Arms: Part B - GB1211 (200 or 100 mg BID) or Placebo in addition to atezolizumab; Part C - Extension of GB1211 (200 or 100 mg BID) or Placebo in addition to atezolizumab
Drug: Atezolizumab — Atezolizumab is an PD-L1 inhibitor administered as an intravenous infusion every three weeks at a dose of 1200mg

SUMMARY:
This study is an open label study followed by a randomised, double-blind, placebo-controlled, parallel group and an extension study to investigate the safety and efficacy of GB1211 (a galectin-3 inhibitor) in combination with atezolizumab in patients with Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
The study will be carried out in three parts: The core study is comprised of part A (dose finding and safety) and part B (efficacy and safety). Part C is an extension phase of the core study to collect long-term safety data.

In part A of the study, open-label sentinel dosing will be undertaken to assess safety and tolerability of GB1211 at 200 mg BID and 100 mg BID in combination with atezolizumab including 4 patients in each dose cohort. Patients enrolled in part A may continue treatment with 200 mg GB1211 BID or 100 mg GB1211 BID and atezolizumab for 12 weeks, after which the patients will be offered treatment in the part C study, if they have achieved clinical benefit as best response during the first 12 weeks of treatment (SD or better response according to RECIST 1.1).

In part B of the study, patients will randomised (1:1) for blinded treatment to receive either GB1211 (200 or 100 mg BID to be selected from part A) or placebo, in addition to atezolizumab, for 12 weeks, after which the patients will be offered treatment in part C, if they have achieved clinical benefit as best response during the first 12 weeks of treatment (SD or better response according to RECIST 1.1).

In part C, this treatment will be blinded until part B has been unblinded. After unblinding, patients will continue to receive the same treatment they had received in part B: GB1211 and atezolizumab or atezolizumab only (no placebo) if they experience continued benefit from treatment. The patients will be treated until disease progression or unacceptable toxicity.

After the end of the study treatment all patients will be followed 4 weeks for safety, regardless of the study part in which the last study treatment was given.

ELIGIBILITY:
Inclusion criteria:

Patients must meet the following criteria for study entry:

1. Must be ≥ 18 years of age at the time of signing the Informed Consent Form (ICF).
2. Must provide signed ICF.
3. Must have the ability to comply with the study protocol, in the investigator's judgment.
4. Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agree to refrain from donating eggs.
5. Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agree to refrain from donating sperm.
6. Diagnosed NSCLC stage IIIB that either progressed after curative therapy (chemoradiation and/or surgery) or is not candidate to curative therapy, or Stage IV metastatic disease (de novo or distant relapse) [According to UICC TNM edition 8].
7. Measurable disease, as defined by RECIST v1.1.
8. Expressing PD-L1 on at least 50% of tumour cells (PD-L1 stained ≥ 50% of tumour cells [TC ≥ 50%] or PD-L1 stained tumour-infiltrating immune cells [IC] covering ≥ 10% of the tumour area [IC ≥ 10%]), as determined through use of the Dako PD-L1 IHC 22C3 pharmDx assay or the Ventana PD-L1 IHC SP263 assay.
9. Agree to have a tumour biopsy that is eligible for Gal-3 expression evaluation before the first study drug dose.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
11. Have not received prior systemic chemotherapy for the treatment of recurrent, advanced or metastatic disease, treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 4 weeks prior to diagnosis of recurrent advanced or metastatic disease.
12. Patients must not have received immune checkpoint inhibitors (ICI) previously.
13. Must be eligible for atezolizumab at 1200 mg every 3 weeks as defined in the atezolizumab product label.
14. Patients receiving therapeutic anticoagulation must be on stable regimen.
15. Adequate haematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    * Absolute neutrophil count (ANC) ≥1.5 x 109/L (1500/µL) without granulocyte colony-stimulating factor support.
    * Lymphocyte count ≥0.5 x 109/L (500/µL).
    * Platelet count ≥ 100 x 109/L (100,000/µL) without transfusion.
    * Haemoglobin ≥ 90 g/L (9 g/dL). Patients may be transfused to meet this criterion.
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions:

      * Patients with documented liver metastases: AST and ALT ≤ 5 x ULN.
      * Patients with documented liver or bone metastases: ALP ≤ 5 x ULN.
    * Total bilirubin ≤ 1.5 x ULN with the following exception:

Patients with known Gilbert disease: total bilirubin ≤ 3 x ULN.

* Creatinine clearance ≥50 mL/min (calculated using the Cockcroft-Gault formula).
* Albumin ≥25 g/L (2.5 g/dL).
* For patients not receiving therapeutic anticoagulation: INR and a PTT ≤1.5 x ULN.

Exclusion criteria:

Patients who meet any of the following criteria will be excluded from study participation.

1. Known contraindications for treatment with PD-1/PD-L1 inhibitors.
2. Patients with known hypersensitivity to GB1211 or any of the excipients.
3. Women who are pregnant or breast-feeding or intending to become pregnant during study treatment or within 9 months after the final dose of study treatment.
4. Women of childbearing potential without a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
5. Women of child-bearing potential or men who are unwilling to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures during the study, and do not agree to refrain from donating sperm or egg cells from the first dose of study drug up to 9 months after the last dose of study drug.
6. Life expectancy ≤ 12 weeks from the expected start of study treatment date.
7. Patients who, in the opinion of the investigator (or designee), should not participate in this study.
8. Patients who participated in a clinical research study involving a new chemical entity or an experimental drug ≤ 4 weeks or 5 half-lives before the first dose of study drug.
9. Presence of oncogenes EGFR (exon 19 deletions, pL858R point mutation in exon 21), or ALK rearrangements.
10. Hepatic impairment of Child Pugh B or C.
11. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test result at screening) and/or hepatitis C virus (HCV).
12. Patients with active human immunodeficiency virus (HIV).
13. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area.
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
14. Patients with severe infection within 4 weeks prior to initiation of study treatment.
15. Patients with acute neurological events (e.g., intracranial or subarachnoid haemorrhage, stroke, intracranial trauma) within 6 months of inclusion.
16. Patients with symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. A CT (with contrast if not contraindicated) or MRI scan of the head must be done at screening to evaluate CNS metastasis in all patients. An MRI scan of the brain is required to confirm or refute the diagnosis of CNS metastases at baseline in the event of an equivocal scan.
17. No tumour specimen, obtained in the last 6 months, is available to analyse galectin expression and it is not feasible to obtain a new specimen (note: cytology samples are admissible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
PART A - To assess the safety and tolerability of GB1211 in combination with atezolizumab. | 3 weeks
  Incidence and severity of adverse events as reported by investigators.
PART B - To assess the safety and tolerability of GB1211 in combination with atezolizumab compared to atezolizumab and placebo | 12 weeks
  Incidence and severity of adverse events
Part B -To assess the efficacy of GB1211 compared to placebo by measuring the change of the longest diameters of target lesions at week 12. | 12 weeks
  Independent central review of CT, PET/CT or MRI scan according to RECIST 1.1
Part C - To assess the long-term safety and tolerability of GB1211 in combination with atezolizumab compared to atezolizumab alone. | 12 - 40 weeks
  Incidence and severity of adverse events.

SECONDARY OUTCOMES:
Part A -To determine the recommended dose (200 mg BID or 100 mg BID) of GB1211 in combination with atezolizumab. | 3 weeks
  Incidence and severity of adverse events as reported by investigators.
Part A and B - To assess response rate according to RECIST v1.1 of GB1211 versus placebo in combination with atezolizumab. | 12 weeks
  Independent central review of CT, PET/CT or MRI scan according to RECIST 1.1
To measure the maximum plasma concentration of GB1211 (Cmax) | 12 weeks
  Plasma concentrations of GB1211 [Time Frame: Part A - Cycle 1 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 2 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 3 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose. Part B - Cycle 1 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose] for the calculation of pharmacokinetic parameter maximum plasma concentration (Cmax) of GB1211
To measure the time of maximum plasma concentration of GB1211 (Tmax) | 12 weeks
  Plasma concentrations of GB1211 [Time Frame: Part A - Cycle 1 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 2 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 3 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose. Part B - Cycle 1 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose] for the calculation of pharmacokinetic parameter time of the maximum plasma concentration (Tmax) of GB1211
To measure the area under the concentration-time curve of GB1211 (AUC) | 12 weeks
  Plasma concentrations of GB1211 [Time Frame: Part A - Cycle 1 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 2 Day 1: pre-dose, 2, 4, 6, 8, 12 hours post-dose; Cycle 3 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose. Part B - Cycle 1 Day 1: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose; End of Treatment: pre-dose, between 2 and 4 hours post-dose, between 4 and 8 hours post-dose] for the calculation of pharmacokinetic parameter area under the plasma concentration versus time curve (AUC) of GB1211
Part C - To assess response rates for those patients who enter the study with at least Stable Disease as best response. | 12 - 40 weeks
  Independent central review of CT, PET/CT or MRI scan according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Francois Ghiringhelli, MD, Principal Investigator — Centre Georges Grancois Leclerc, Dijon
Locations (5):
- France (2):
  - Centre Georges Grancois Leclerc, Dijon
  - CHRU, Tours
- Samodzielny Publiczny Zespol Gruzlicy I Chorob Pluc, Olsztyn, Poland
- Spain (2):
  - Hospital Universitario y Politécnico La Fe, Valencia, València
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No